## **Informed Consent Form**

Title: Well-Child Visit Video Project

Date: 03/23/2021

NCT#: NCT05011292

Study Title: Well-Child Visit Video Project

IRB #: STUDY00001393

Principal Investigator: Jean Welsh, PhD, MPH, RN, Emory School of Medicine, Department of Pediatrics

<u>Funding Source:</u> The Global Center for Diabetes Translation Research, pilot grant program.

## **Introduction and Study Overview**

A few of the doctors here at Hughes Spalding are working with researchers at Emory University to do a study to see if using videos as part of well-child visits is a good way for doctors to share important information about infant feeding with parents. We would like to invite you to be a part of this study. Participating involves:

- 1. Watching a video today and completing a set of questions before and after it: 6-7 minutes
- 2. Completing a short survey about infant feeding if you return to the clinic for your child's next scheduled well-child visit: 2 minutes
- 3. Completing a follow-up survey by email or text four to five months from now: 5 minutes

... for a total of about 20 minutes. Those who participate will be sent, a \$20 gift card by email or text after completing the follow-up survey. Whether or not you decide to participate is your choice. If you decide not to, it won't have any effect on the care provided to your child by the clinic team. If you decide to participate now, and change your mind later, you can stop any time.

Possible risks to the study include loss of confidentiality and the time lost completing the surveys. The risk of loss of confidentiality will be kept low by using study numbers instead of names and saving identifying information on password protected computers, to which only select study staff will have access. There is no direct benefit to you or your child if you participate and no risk if you do not. We hope that the information collected will benefit parents and children in the future.

Study records can be opened by court order. They also may be provided in response to a subpoena or a request for the production of documents. Certain offices and people other than the researchers may look at study records. Government agencies, Emory employees and Children's employees overseeing proper study conduct may look at your study records. These offices include the Office for Human Research Protections, the funder, the Emory and Children's Institutional Review Boards, and the Emory and Children's Offices of Research Compliance. Study funders may also look at your study records. Emory will keep any research records we create private to the extent we are required to do so by law. Other than as a result of a court order, your data from this study will not be shared with anyone outside of this study. A description of this clinical trial will be available on http://www.ClinicalTrials.gov. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time

## **Contact Information**

| If you have questions about this study, your part in it, or | if you have questions, or concerns about the research you may |
|---|---|
| contact the following: | |
| Jean Welsh, Principal Investigator: | |

If you have questions about your rights at research participant, complaints about the research or an issue you rather discuss with someone outside the research team, contact the Emory Institutional Review Board at